CLINICAL TRIAL: NCT03499470
Title: The Effectiveness of Structured Discharge and Follow-up Protocol on Readmission Rate in COPD Patients Receiving LTOT and NIV: A Multicenter Randomized Trial
Brief Title: Structured Discharge and Follow-up Protocol for COPD Patients Receiving LTOT and NIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: Celal Bayar University (Other); Ege University (Other); Gazi University (Other); Duzce University (Other); Cukurova University (Other); Ataturk University (Other); Uludag University (Other); Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other); Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other); Ordu University (Other); Hacettepe University (Other); Turkish Directorate General of Public Health (Unknown); Istanbul University - Cerrahpasa (Other); Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Begum Ergan, Instructor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20.478.486.359
Record Dates: First submitted 2018-04-02; First posted 2018-04-17 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: COPD Exacerbation; Noninvasive Ventilation; Long Term Oxygen Therapy; Chronic Respiratory Failure
Keywords: copd; exacerbation; structured discharge; readmission; chronic respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention mainly consists of a developed protocol for education about the disease and medications AND an education of the equipment and how to use it to have the best benefit.
  Actions in structured discharge and follow up protocol:
  1. Patient education for disease severity and medications
  2. Education of family/relatives about medications and types of equipment
  3. Detailed education for LTOT and/or NIV (how to use, duration of use, solutions for possible common problems)
  4. Preparation of home environment for patients needs
  5. Regular telephone visits on day 7 and day 14 after discharge and telephone visits in emergency situations and early referral to the hospital when needed
  6. Outpatient control for the first month
  Interventions: Other: Protocol for structured discharge and follow-up
- Control (No Intervention): Control patients will receive usual care

INTERVENTIONS:
Other: Protocol for structured discharge and follow-up
  Arms: Intervention

SUMMARY:
Readmission to hospital is one of the most important problems in chronic obstructive pulmonary disease (COPD) patients who developed chronic respiratory failure. Patients receiving long-term oxygen therapy (LTOT) and noninvasive ventilation (NIV) constitute the most vulnerable group because of the need for comprehensive care. However, because of lack of health care support systems in Turkey, many advanced COPD patients are hospitalized due to preventable problems such as insufficient knowledge about the therapies, nonadherence to therapy and technical issues related to LTOT/NIV equipment. The aim of this multicenter randomized trial is to find out whether a structured discharge and follow-up protocol reduce the rate of unplanned, COPD-related hospital readmissions over 90 days in patients receiving LTOT or NIV.

DETAILED DESCRIPTION:
The study is planned with Turkish Thoracic Society and Global Alliance Against Respiratory Disease-Turkey partnership and being carried out 10 centers throughout Turkey. COPD patients who are prescribed long-term oxygen therapy for hypoxemic respiratory failure and/or noninvasive ventilation for hypercapnic respiratory failure will be included in the study and will be randomized to either intervention or control arm. The intervention mainly consists of not only education about the disease and medications but also the education of the equipment and how to use it to have the best benefit. Control arm patients will receive usual care, which consists of basic education of the patient about the therapies. The primary outcome of the study is readmission in 90 days.

ELIGIBILITY:
Inclusion Criteria:

COPD patients who developed chronic respiratory failure and are eligible for long-term oxygen therapy (LTOT) or noninvasive ventilation (NIV) according to Turkish National Social Security regulations

Definitions:

COPD: The diagnosis of COPD is made according to GOLD criteria Chronic respiratory failure: PaO2>60mmHg at room air and/or PaCO2> 45

Eligibility for LTOT:

1. PaO2 ≤ 55 mmHg or SaO2 ≤ 88% under room air
2. PaO2 value of 55-59 mmHg or SaO2 ≤ 89% and cor pulmonale with hematocrit >55 or p pulmonale in ECG or congestive heart failure.

Eligibility for NIV:

1. PaCO2≥55 mmHg or
2. PaCO2 50 to 54 mmHg and nocturnal desaturation ≤ %88 for 5 minutes under 2lt/min nasal O2 therapy 3. PaCO2 50 to 54 mmHg and >2 exacerbations within the last year

Exclusion Criteria:

1. Patients receiving LTOT or NIV for a different cause 2. Patients who do not give consent 3. Patients who are unable to be followed up regularly due to reasons such as living far from study center, lack of family support, unwillingness or inability to contact regularly.

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Readmission rate | 90days
  The rate of unplanned, COPD-related hospital readmissions over 90 days after discharge

SECONDARY OUTCOMES:
Time to first exacerbation | 90 days
  Time to first exacerbation after discharge
Rate of exacerbation | 90 days
  Total COPD exacerbation rate within 90 days after discharge
Rate of hospitalization | 90 days
  Total hospitalization number due to COPD within 90 days after discharge
Compliance to treatment | 90 days
  Compliance to LTOT and NIV therapies will be assessed by duration of use (number of hours per day and number of nights per week) within 90 days after discharge.
Long term survival | One year
  One year survival after discharge

CONTACTS AND LOCATIONS:
Overall Officials: BEGUM ERGAN, MD, Study Director — Dokuz Eylul University; TUGBA GOKTALAY, MD, Study Director — Celal Bayar University; PINAR ERGUN, MD, Principal Investigator — Health Sciences University Ataturk Chest Diseases and Chest Surgery Hospital; ALEV GURGUN, MD, Principal Investigator — Ege University; METIN AKGUN, MD, Principal Investigator — Ataturk University; NURDAN KOKTURK, MD, Principal Investigator — Gazi University; EZGI OZYILMAZ, MD, Principal Investigator — Cukurova University; ASLI DILEKTASLI, MD, Principal Investigator — Uludag University; BIRSEN OCAKLI, MD, Principal Investigator — Health Sciences University Sureyyapasa Chest Diseases and Chest Surgery Hospital; ONER BALBAY, MD, Principal Investigator — Duzce University
Locations (10):
- Turkey (Türkiye) (10):
  - Dokuz Eylul University, Izmir, Narlıdere
  - Cukurova University, Adana
  - Gazi University, Ankara
  - Health Sciences University Ataturk Chest Diseases and Chest Surgery Hospital, Ankara
  - Uludag University, Bursa
  - Duzce University, Düzce
  - Ataturk University, Erzurum
  - Health Sciences University Sureyyapasa Chest Diseases and Chest Surgery Hospital, Istanbul
  - Ege University, Izmir
  - Celal Bayar University, Manisa